CLINICAL TRIAL: NCT07215273
Title: A Phase 2, Multicenter, Randomized, Double-blind Study of Safety and Efficacy of EL219 Versus Standard of Care (Liposomal Amphotericin B Followed by Voriconazole) for Early Antifungal Therapy of Suspected Invasive Mould Infections
Brief Title: Study of EL219 vs Standard of Care for Early Antifungal Therapy of Suspected Invasive Mould Infections
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Elion Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EL219.IV.2.04
Record Dates: First submitted 2025-09-24; First posted 2025-10-10 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Suspected Invasive Mould Infection
Keywords: Invasive Mould Infection; Mould infection; Prophylaxis for Invasive Mould Infection; Anti-fungal therapy; Invasive Mold Infection; Mold infection; Prophylaxis for Invasive Mold Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EL219 (Experimental): Participants randomized to EL219 will receive a single loading dose of EL219 at 2 mg/kg via IV infusion on Day 1, and 1.5 mg/kg IV infusions on Days 8, 15, 22, 29, and 36.
  To maintain the blind, placebo IV infusions will be administered on Days 2-7 and 9-14 corresponding to Liposomal Amphotericin B (LAmB) dosing; thereafter, twice daily oral or IV placebo will be administered corresponding to voriconazole dosing until Day 42/EOT.
  Interventions: Drug: EL219
- Antifungal Comparator (Active Comparator): Standard of Care- Participants will receive LAmB 3 mg/kg IV infusions for at least 14 days and up to 42 days.Voriconazole Daily Dosing- Loading 6 mg/kg via IV infusion every 12 hrs for the first 24 hrs. Post-loading: 4 mg/kg oral every 12 hrs (admin as 50 mg overencapsulated tabs) OR 4 mg/kg via IV infusion every 12 hrs
  Participants on oral therapy will be administered placebo IV infusions corresponding to EL219 on Days 15, 22, 29, and 36 to maintain the blind. Participants may switch from LAmB to voriconazole (oral or IV) at any time, if any of the following occur:
  * Dx. of proven or probable IA per EORTC/MSG criteria
  * Other proven or probable susceptible MI
  * Possible IMI that requires continued antifungal therapy
  * Toxicity: Acute renal injury, hypokalemia or hypomagnesemia uncontrolled with IV supplementation, Increase in ALT to 3× baseline and/or total serum bilirubin 3× baseline, Intractable IRR
  * Change to oral due to imminent hosp. discharge
  Interventions: Drug: Antifungal Comparator

INTERVENTIONS:
Drug: EL219 — EL219 is specifically being developed for early antifungal therapy (EAT), when infection is suspected due to highly suggestive signs and symptoms of disease; in high-risk people, antifungals are recommended even before confirmation of the microbial cause of infection, because delayed therapy is associated with poor outcomes in those who lack adequate immune responses. EL219 may provide a once-weekly alternative to LAmB and other polyenes that could also reduce the toxicities that often limit the frequency and duration of administration for these highly efficacious antifungals.
  Arms: EL219
Drug: Antifungal Comparator — Placebo IV infusions (inf.) on Days 2-7, 9-14 to match LAmB dosing. Thereafter, twice daily oral or IV placebo equal to voriconazole dosing until Day 42/EOT. Active Comparator/SoC will receive LAmB 3 mg/kg IV inf. for at least 14 days & up to 42 days. Voriconazole daily dosing loading 6 mg/kg via IV inf. every 12hrs for first 24hrs. Post-load: 4 mg/kg oral every 12hrs (50 mg tablets) or 4 mg/kg via IV inf. every 12hrs. Oral therapy will be admin., placebo IV inf. to match EL219 on Days 15, 22, 29 & 36. May switch from LAmB to voriconazole (oral or IV) if any of these occur: diagnosis of proven or probable IA per EORTC/MSG criteria, other proven or probable susceptible mould infection, possible IMI requiring continued antifungal therapy. Toxicity: acute renal injury, hypokalemia or hypomagnesemia not controlled by IV supplementation, increase ALT 3×baseline and/or total serum bilirubin 3×baseline, intractable IRR. Need to switch to oral therapy for imminent hospital discharge.
  Arms: Antifungal Comparator

SUMMARY:
The purpose of this study is to determine if EL219 is safe and effective compared to the standard of care for early treatment of suspected invasive mould infection.

DETAILED DESCRIPTION:
A Phase 2, multicenter, randomized, double-blind Study of Safety and Efficacy of EL219 versus standard anti-fungal therapy for suspected Invasive Mould Infections.

ELIGIBILITY:
Inclusion Criteria:

Participants who meet ALL the following inclusion criteria will be eligible to participate in the study:

1. Willing and able to provide written informed consent.
2. Males or females 18 years and older,
3. Are at risk for invasive fungal infections (IFIs), with one of the following:

   1. Receipt of a bone marrow transplant (BMT) from an allogeneic donor, with blood, bone marrow, or cord blood as stem cell source.
   2. Receiving or have recently (within 1 month) received cytotoxic, biologic, or immune modulating therapy(ies) for hematological malignancy.
   3. Receipt of corticosteroids at mean minimum doses of 0.3 mg/kg/day prednisone equivalent for more than 3 weeks.
   4. Receipt of other recognized T-cell immunosuppressants, such as cyclosporin, tumor necrosis factor alpha (TNF-α) blockers, or specific monoclonal antibodies during the last 3 months.
   5. Inherited severe immunodeficiency

Has suspected invasive mould infection (IMI) as defined by one or both of the following:

1. Results of an assay having regulatory clearance in Europe or the United States (Conformité Européene [CE] mark or United States Food and Drug Administration [US FDA] 510k clearance), demonstrating positivity at validated cut-off that is suggestive of IMI, but does not meet microbiologic criteria for probable invasive aspergillosis (IA; as defined by European Organization for Research and Treatment of Cancer/Invasive Fungal Infections Cooperative Group and the National Institute of Allergy and Infectious Diseases Mycoses Study Group [EORTC/MSG]). Diagnostic tests must have regulatory approval in the region in which the diagnostic is performed and are inclusive of Platelia serum galactomannan, serum or bronchoalveolar lavage (BAL) polymerase chain reaction (PCR), serum or BAL Aspergillus antigen lateral flow assays (LFAs; IMMY, OLM Diagnostics, or TECO®), or urine MycoMEIA®-Aspergillus assay
2. Abnormal findings on chest computed tomography (CT) scan without alternative microbiologic diagnosis Note: If CT of the chest is used to establish eligibility it must be performed within 7 days prior to randomization.

   5. Must have IV access in place or to be placed prior to beginning IV study therapy.

   6. Must be willing to adhere to dosing, study visit schedule, and mandatory diagnostic procedures.

   7. Female participants must meet 1 of the following criteria: A woman of childbearing potential (WOCBP) must agree to use a highly effective, preferably user-independent method of contraception (failure rate of <1% per year when used consistently and correctly) for at least 30 days prior to screening and agree to remain on a highly effective method until 2 months after study drug administration.

   8. A WOCBP must have a negative highly sensitive serum pregnancy test (β-human chorionic gonadotropin) at screening and a negative urine pregnancy test on Day -1 before study drug administration.

   9. Females must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for a period of at least 2 months after study drug administration.

   10. Male participants must be vasectomized or agree to abstain from intercourse or if engaging in sexual activity that has risk of pregnancy, must agree to use a double barrier method and agree not to donate sperm during the study and for at least 120 days after study drug administration.

Exclusion Criteria:

Participants must NOT meet any of the following exclusion criteria:

1. Diagnosis of proven or probable IMI within 1 month prior to randomization (including meeting the criteria for proven or probable IMI during the screening period), or relapsed/recurrent IMI which has not responded to other antifungal therapies.

2. Participant has received prior antifungal treatment (azole prophylaxis permitted) for >96 hours prior to randomization.

3. Systemic bacterial infection diagnosed within the 14 days prior to randomization.

4. Participants with 1 or more of the following laboratory abnormalities as defined by the National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE) v5.0:

1. Alanine aminotransferase (ALT) ≥5 × upper limit of normal (ULN).
2. Total serum bilirubin ≥5 × ULN (excluding Gilbert's Syndrome).
3. Serum creatinine ≥2 mg/dL or creatinine clearance (CrCL) ≤30 mL/minute. 5. Known cirrhosis of the liver, diagnosed according to country or Medical Society-specific guidelines and documented in the medical records prior to screening.

   6. Diagnosed symptomatic heart failure with left ventricular ejection fraction (LVEF) at rest ≤50%, or shortening fraction ≤26%.

   Diagnosed reduced lung function with either diffusion capacity (corrected for hemoglobin) or forced expiratory volume in 1 second (FEV1) ≤65% of predicted value, or oxygen (O2) saturation ≤82% on room air.

   8. Receiving either hemodialysis or peritoneal dialysis. 9. Personal or family history of long QT interval on ECG (QT) syndrome or a prolonged QT interval corrected for heart rate by Fridericia's formula (QTcF; >470 msec in males and >480 msec in females).

   10. Current or projected use of the following medications or drug classes known to interact with voriconazole: terfenadine, astemizole, cisapride, pimozide, quinidine, sirlolimus, rifampin, phenytoin, carbamazepine, ritonavir or other protease inhibitors, efavirenz or other non-nucleoside reductase inhibitors, rifabutin, St. John's Wort, ergot alkaloids, or long-acting barbiturates.

   11. History of hereditary problems with galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption.

   12. Known hypersensitivity to EL219 Powder for Injection, LAmB®, voriconazole, other azole antifungal, or any of their excipients.

   13. History of severe allergic response to mRNA-based severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) vaccine and/or polyethylene glycol (PEG)-containing products.

   14. Previous participation in any study using an investigational drug within 28 days of study drug administration on Day 1 or 5 half-lives of the drug, whichever is longer, and throughout the study until the Day 56 Safety Follow-up visit is completed. Concurrent participation in another trial may be allowed (e.g., interventional trial with a previously approved study drug[s] or observational trial). In such cases, Sponsor Medical Monitor should be consulted prior to enrolling a potential participant.

   15. Prior recipient of orthotopic lung transplant. 16. Likely to transition to hospice care for underlying hematological malignancy, is under a Do Not Resuscitate (DNR) order, or is receiving best supportive care only.

   17. Female participants who are pregnant or lactating or planning to become pregnant within 2 months following study drug administration.

   18. The Principal Investigator (PI) determines the participant should not participate in the study.

   19. Considered unlikely to follow up for required days due to logistic concerns (i.e., home location relative to study site).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome/Measure All-Cause Mortality | From enrollment to the end of treatment at Day 42
  All-cause mortality at Day 42 in the Intent-to-Treat (ITT) analysis set.
Primary Outcome/Measure SAE TEAE | From enrollment to the end of treatment at Day 42
  Serious adverse events and treatment-emergent adverse events categorized in a tiered approach in the Safety analysis set.

SECONDARY OUTCOMES:
Secondary Outcome Measure-Overall Success | From enrollment through Day 42
  Overall success at Day 42, confirmed by the Data Review Committee, in the population with proven or probable IA (modified Intent-to-Treat)
Secondary Outcome Measure-Participant is Alive | From enrollment through Day 42
  Participant is alive, favorable composite clinical, mycologic, and radiographic response (European Organization for Research and Treatment of Cancer/Invasive Fungal Infections Cooperative Group and the National Institute of Allergy and Infectious Diseases Mycoses Study Group criteria)
Secondary Outcome Measure-EAT Success | From enrollment through Day 42
  Early antifungal therapy (EAT) success at Day 42 in the ITT analysis set defined by non-occurrence of the following: death, receipt of non-study drug systemic antifungal therapy for a cumulative exposure >10 days for progression of disease and/or toxicity, missing data (classified as indeterminate but analyzed as a failure).
Secondary Outcome Measure- Breakthrough | From enrollment through Day 14
  Breakthrough possible, probable, or proven IFI established after 14 days of study drug in the ITT analysis set
Secondary Outcome Measure- Hospitalization | From enrollment through Day 42
  Duration of the initial hospitalization after randomization, in the ITT analysis set
Secondary Outcome Measure-Rehospitalization | From enrollment through Day 42
  Reason for and duration of rehospitalization after discharge from the initial hospitalization in the ITT analysis set.

CONTACTS AND LOCATIONS:
Overall Officials: Taylor G. Sandison, MD, Study Director — Sponsor: Elion Therapeutics, Chief Medical Officer
Locations (2):
- United States (2):
  - Washington U., St Louis, Missouri
  - U. of Texas, MD Anderson, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.

REFERENCES:
- [Background] Adler-Moore J, Lewis RE, Bruggemann RJM, Rijnders BJA, Groll AH, Walsh TJ. Preclinical Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Antifungal Activity of Liposomal Amphotericin B. Clin Infect Dis. 2019 May 2;68(Suppl 4):S244-S259. doi: 10.1093/cid/ciz064. PMID 31222254
- [Background] AmBisome® (amphotericin B) liposome for injection [Prescribing Information]. Foster City, CA: Gilead Sciences, Inc.; 2022.
- [Background] AmBisome Liposomal 50 mg Powder for dispersion for infusion [Summary of Product Characteristics]. Foster City, CA: Gilead Sciences, Inc.; May 2024.
- [Background] Anderson TM, Clay MC, Cioffi AG, Diaz KA, Hisao GS, Tuttle MD, Nieuwkoop AJ, Comellas G, Maryum N, Wang S, Uno BE, Wildeman EL, Gonen T, Rienstra CM, Burke MD. Amphotericin forms an extramembranous and fungicidal sterol sponge. Nat Chem Biol. 2014 May;10(5):400-6. doi: 10.1038/nchembio.1496. Epub 2014 Mar 30. PMID 24681535
- [Background] Bowden R, Chandrasekar P, White MH, Li X, Pietrelli L, Gurwith M, van Burik JA, Laverdiere M, Safrin S, Wingard JR. A double-blind, randomized, controlled trial of amphotericin B colloidal dispersion versus amphotericin B for treatment of invasive aspergillosis in immunocompromised patients. Clin Infect Dis. 2002 Aug 15;35(4):359-66. doi: 10.1086/341401. Epub 2002 Jul 25. PMID 12145716
- [Background] Burke MD, He X, Cook C, Petrov GA, Long S, Coffin MD. Stability enhancement of drug layered pellets in a fixed dose combination tablet. AAPS PharmSciTech. 2013 Mar;14(1):312-20. doi: 10.1208/s12249-012-9911-3. Epub 2013 Jan 15. PMID 23319298
- [Background] Chamilos G, Luna M, Lewis RE, Chemaly R, Raad II, Kontoyiannis DP. Effects of liposomal amphotericin B versus an amphotericin B lipid complex on liver histopathology in patients with hematologic malignancies and invasive fungal infections: a retrospective, nonrandomized autopsy study. Clin Ther. 2007 Sep;29(9):1980-6. doi: 10.1016/j.clinthera.2007.09.016. PMID 18035197
- [Background] Cornely OA, Maertens J, Bresnik M, Ebrahimi R, Dellow E, Herbrecht R, Donnelly JP. Efficacy outcomes in a randomised trial of liposomal amphotericin B based on revised EORTC/MSG 2008 definitions of invasive mould disease. Mycoses. 2011 Sep;54(5):e449-55. doi: 10.1111/j.1439-0507.2010.01947.x. Epub 2010 Oct 11. PMID 21039936
- [Background] Cornely OA, Maertens J, Bresnik M, Ebrahimi R, Ullmann AJ, Bouza E, Heussel CP, Lortholary O, Rieger C, Boehme A, Aoun M, Horst HA, Thiebaut A, Ruhnke M, Reichert D, Vianelli N, Krause SW, Olavarria E, Herbrecht R; AmBiLoad Trial Study Group. Liposomal amphotericin B as initial therapy for invasive mold infection: a randomized trial comparing a high-loading dose regimen with standard dosing (AmBiLoad trial). Clin Infect Dis. 2007 May 15;44(10):1289-97. doi: 10.1086/514341. Epub 2007 Apr 9. PMID 17443465
- [Background] Davis SA, Vincent BM, Endo MM, Whitesell L, Marchillo K, Andes DR, Lindquist S, Burke MD. Nontoxic antimicrobials that evade drug resistance. Nat Chem Biol. 2015 Jul;11(7):481-7. doi: 10.1038/nchembio.1821. Epub 2015 Jun 1. PMID 26030729
- [Background] Donnelly JP, Chen SC, Kauffman CA, Steinbach WJ, Baddley JW, Verweij PE, Clancy CJ, Wingard JR, Lockhart SR, Groll AH, Sorrell TC, Bassetti M, Akan H, Alexander BD, Andes D, Azoulay E, Bialek R, Bradsher RW, Bretagne S, Calandra T, Caliendo AM, Castagnola E, Cruciani M, Cuenca-Estrella M, Decker CF, Desai SR, Fisher B, Harrison T, Heussel CP, Jensen HE, Kibbler CC, Kontoyiannis DP, Kullberg BJ, Lagrou K, Lamoth F, Lehrnbecher T, Loeffler J, Lortholary O, Maertens J, Marchetti O, Marr KA, Masur H, Meis JF, Morrisey CO, Nucci M, Ostrosky-Zeichner L, Pagano L, Patterson TF, Perfect JR, Racil Z, Roilides E, Ruhnke M, Prokop CS, Shoham S, Slavin MA, Stevens DA, Thompson GR, Vazquez JA, Viscoli C, Walsh TJ, Warris A, Wheat LJ, White PL, Zaoutis TE, Pappas PG. Revision and Update of the Consensus Definitions of Invasive Fungal Disease From the European Organization for Research and Treatment of Cancer and the Mycoses Study Group Education and Research Consortium. Clin Infect Dis. 2020 Sep 12;71(6):1367-1376. doi: 10.1093/cid/ciz1008. PMID 31802125
- [Background] Empiric antifungal therapy in febrile granulocytopenic patients. EORTC International Antimicrobial Therapy Cooperative Group. Am J Med. 1989 Jun;86(6 Pt 1):668-72. doi: 10.1016/0002-9343(89)90441-5. PMID 2658574
- [Background] European Medicines Agency. Good practice guide on recording, coding, reporting, and assessment of medication errors (EMA/762563/2014). 2015.
- [Background] Clinical Trials Regulation (EU) No. 536/2014 of the European Parliament and the Council of 16 April 2014 on Clinical Trials on Medicinal Products for Human Use, and Repealing Directive 2001/20/EC Text with EEA relevance - Annex III.
- [Background] Fiorcari S, Maffei R, Vallerini D, Scarfo L, Barozzi P, Maccaferri M, Potenza L, Ghia P, Luppi M, Marasca R. BTK Inhibition Impairs the Innate Response Against Fungal Infection in Patients With Chronic Lymphocytic Leukemia. Front Immunol. 2020 Aug 28;11:2158. doi: 10.3389/fimmu.2020.02158. eCollection 2020. PMID 32983178
- [Background] Fleming RV, Kantarjian HM, Husni R, Rolston K, Lim J, Raad I, Pierce S, Cortes J, Estey E. Comparison of amphotericin B lipid complex (ABLC) vs. ambisome in the treatment of suspected or documented fungal infections in patients with leukemia. Leuk Lymphoma. 2001 Feb;40(5-6):511-20. doi: 10.3109/10428190109097650. PMID 11426524
- [Background] Garbuzenko O, Zalipsky S, Qazen M, Barenholz Y. Electrostatics of PEGylated micelles and liposomes containing charged and neutral lipopolymers. Langmuir. 2005 Mar 15;21(6):2560-8. doi: 10.1021/la0479105. PMID 15752053
- [Background] Gillis EP, Burke MD. A simple and modular strategy for small molecule synthesis: iterative Suzuki-Miyaura coupling of B-protected haloboronic acid building blocks. J Am Chem Soc. 2007 May 30;129(21):6716-7. doi: 10.1021/ja0716204. Epub 2007 May 9. No abstract available. PMID 17488084
- [Background] Girmenia C, Aversa F, Busca A, Candoni A, Cesaro S, Luppi M, Pagano L, Rossi G, Venditti A, Nosari AM; Sorveglianza Epidemiologica delle Infezioni Fungine nelle Emopatie Maligne; Invasive Fungal Infections Cooperative Group of the European Organization for Research and Treatment of Cancer; Gruppo Italiano Malattie Ematologiche dell'Adulto; Associazione Italiana Ematologia ed Oncologia Pediatrica; Gruppo Italiano Trapianto di Midollo Osseo. A hematology consensus agreement on antifungal strategies for neutropenic patients with hematological malignancies and stem cell transplant recipients. Gruppo Italiano Malattie Ematologiche dell'Adulto, Gruppo Italiano Trapianto di Midollo Osseo, Associazione Italiana Ematologia ed Oncologia Pediatrica, Invasive Fungal Infections Cooperative Group of the European Organization for Research and Treatment of Cancer and Sorveglianza Epidemiologica delle Infezioni Fungine nelle Emopatie Maligne. Hematol Oncol. 2013 Sep;31(3):117-26. doi: 10.1002/hon.2031. Epub 2012 Oct 5. PMID 23037867
- [Background] Gray KC, Palacios DS, Dailey I, Endo MM, Uno BE, Wilcock BC, Burke MD. Amphotericin primarily kills yeast by simply binding ergosterol. Proc Natl Acad Sci U S A. 2012 Feb 14;109(7):2234-9. doi: 10.1073/pnas.1117280109. Epub 2012 Jan 17. PMID 22308411
- [Background] Hong Y, Ramzan I, McLachlan AJ. Hepatobiliary disposition of liposomal amphotericin B in the isolated perfused rat liver. J Pharm Sci. 2005 Jan;94(1):169-76. doi: 10.1002/jps.20239. PMID 15761940
- [Background] Jarvis JN, Lawrence DS, Meya DB, Kagimu E, Kasibante J, Mpoza E, Rutakingirwa MK, Ssebambulidde K, Tugume L, Rhein J, Boulware DR, Mwandumba HC, Moyo M, Mzinganjira H, Kanyama C, Hosseinipour MC, Chawinga C, Meintjes G, Schutz C, Comins K, Singh A, Muzoora C, Jjunju S, Nuwagira E, Mosepele M, Leeme T, Siamisang K, Ndhlovu CE, Hlupeni A, Mutata C, van Widenfelt E, Chen T, Wang D, Hope W, Boyer-Chammard T, Loyse A, Molloy SF, Youssouf N, Lortholary O, Lalloo DG, Jaffar S, Harrison TS; Ambition Study Group. Single-Dose Liposomal Amphotericin B Treatment for Cryptococcal Meningitis. N Engl J Med. 2022 Mar 24;386(12):1109-1120. doi: 10.1056/NEJMoa2111904. PMID 35320642
- [Background] Lepak AJ, VanScoy B, Rubino C, Ambrose PG, Andes DR. In vivo pharmacodynamic characterization of a next-generation polyene, SF001, in the invasive pulmonary aspergillosis mouse model. Antimicrob Agents Chemother. 2024 Mar 6;68(3):e0163123. doi: 10.1128/aac.01631-23. Epub 2024 Feb 6. PMID 38319077
- [Background] Lewandowska A, Soutar CP, Greenwood AI, Nimerovsky E, De Lio AM, Holler JT, Hisao GS, Khandelwal A, Zhang J, SantaMaria AM, Schwieters CD, Pogorelov TV, Burke MD, Rienstra CM. Fungicidal amphotericin B sponges are assemblies of staggered asymmetric homodimers encasing large void volumes. Nat Struct Mol Biol. 2021 Dec;28(12):972-981. doi: 10.1038/s41594-021-00685-4. Epub 2021 Dec 9. PMID 34887566
- [Background] Miceli MH, Chandrasekar P. Safety and efficacy of liposomal amphotericin B for the empirical therapy of invasive fungal infections in immunocompromised patients. Infect Drug Resist. 2012;5:9-16. doi: 10.2147/IDR.S22587. Epub 2012 Jan 11. PMID 22294858
- [Background] Mohamed M, Abu Lila AS, Shimizu T, Alaaeldin E, Hussein A, Sarhan HA, Szebeni J, Ishida T. PEGylated liposomes: immunological responses. Sci Technol Adv Mater. 2019 Jun 26;20(1):710-724. doi: 10.1080/14686996.2019.1627174. eCollection 2019. PMID 31275462
- [Background] Morelle C, Mukherjee A, Zhang J, Fani F, Khandelwal A, Gingras H, Trottier J, Barbier O, Leprohon P, Burke MD, Ouellette M. Well-Tolerated Amphotericin B Derivatives That Effectively Treat Visceral Leishmaniasis. ACS Infect Dis. 2021 Aug 13;7(8):2472-2482. doi: 10.1021/acsinfecdis.1c00245. Epub 2021 Jul 20. PMID 34282886
- [Background] Nasillo V, Lagreca I, Vallerini D, Barozzi P, Riva G, Maccaferri M, Paolini A, Forghieri F, Fiorcari S, Maffei R, Martinelli S, Atene CG, Castelli I, Marasca R, Potenza L, Comoli P, Manfredini R, Tagliafico E, Trenti T, Luppi M. BTK Inhibitors Impair Platelet-Mediated Antifungal Activity. Cells. 2022 Mar 16;11(6):1003. doi: 10.3390/cells11061003. PMID 35326454
- [Background] Palacios DS, Dailey I, Siebert DM, Wilcock BC, Burke MD. Synthesis-enabled functional group deletions reveal key underpinnings of amphotericin B ion channel and antifungal activities. Proc Natl Acad Sci U S A. 2011 Apr 26;108(17):6733-8. doi: 10.1073/pnas.1015023108. Epub 2011 Feb 28. PMID 21368185
- [Background] Patterson TF, Thompson GR 3rd, Denning DW, Fishman JA, Hadley S, Herbrecht R, Kontoyiannis DP, Marr KA, Morrison VA, Nguyen MH, Segal BH, Steinbach WJ, Stevens DA, Walsh TJ, Wingard JR, Young JA, Bennett JE. Executive Summary: Practice Guidelines for the Diagnosis and Management of Aspergillosis: 2016 Update by the Infectious Diseases Society of America. Clin Infect Dis. 2016 Aug 15;63(4):433-42. doi: 10.1093/cid/ciw444. PMID 27481947
- [Background] Scardina T, Fawcett AJ, Patel SJ. Amphotericin-Associated Infusion-Related Reactions: A Narrative Review of Pre-Medications. Clin Ther. 2021 Oct;43(10):1689-1704. doi: 10.1016/j.clinthera.2021.09.011. Epub 2021 Oct 23. PMID 34696915
- [Background] Segal BH, Almyroudis NG, Battiwalla M, Herbrecht R, Perfect JR, Walsh TJ, Wingard JR. Prevention and early treatment of invasive fungal infection in patients with cancer and neutropenia and in stem cell transplant recipients in the era of newer broad-spectrum antifungal agents and diagnostic adjuncts. Clin Infect Dis. 2007 Feb 1;44(3):402-9. doi: 10.1086/510677. Epub 2007 Jan 2. PMID 17205448
- [Background] Stone NR, Bicanic T, Salim R, Hope W. Liposomal Amphotericin B (AmBisome((R))): A Review of the Pharmacokinetics, Pharmacodynamics, Clinical Experience and Future Directions. Drugs. 2016 Mar;76(4):485-500. doi: 10.1007/s40265-016-0538-7. PMID 26818726
- [Background] Stott KE, Moyo M, Ahmadu A, Kajanga C, Gondwe E, Chimang'anga W, Chasweka M, Leeme TB, Molefi M, Chofle A, Bidwell G, Changalucha J, Unsworth J, Jimenez-Valverde A, Lawrence DS, Mwandumba HC, Lalloo DG, Harrison TS, Jarvis JN, Hope W, Martson AG. Population pharmacokinetics of liposomal amphotericin B in adults with HIV-associated cryptococcal meningoencephalitis. J Antimicrob Chemother. 2022 Dec 23;78(1):276-283. doi: 10.1093/jac/dkac389. PMID 36411251
- [Background] Szebeni J, Simberg D, Gonzalez-Fernandez A, Barenholz Y, Dobrovolskaia MA. Roadmap and strategy for overcoming infusion reactions to nanomedicines. Nat Nanotechnol. 2018 Dec;13(12):1100-1108. doi: 10.1038/s41565-018-0273-1. Epub 2018 Oct 22. PMID 30348955
- [Background] VFEND® (voriconazole) tablets, for oral use; and (voriconazole) for injection, for intravenous use [Prescribing Information]. New York, NY: Roerig Division of Pfizer Inc.; 2019.
- [Background] Voriconazole 50 mg film-coated tablets [Summary of Product Characteristics]. Sandwich, UK: Pfizer Limited; 2025.
- [Background] Vukovic L, Khatib FA, Drake SP, Madriaga A, Brandenburg KS, Kral P, Onyuksel H. Structure and dynamics of highly PEG-ylated sterically stabilized micelles in aqueous media. J Am Chem Soc. 2011 Aug 31;133(34):13481-8. doi: 10.1021/ja204043b. Epub 2011 Aug 9. PMID 21780810
- [Background] Wilcock BC, Endo MM, Uno BE, Burke MD. C2'-OH of amphotericin B plays an important role in binding the primary sterol of human cells but not yeast cells. J Am Chem Soc. 2013 Jun 12;135(23):8488-91. doi: 10.1021/ja403255s. Epub 2013 Jun 3. PMID 23718627
- [Background] Woerly EM, Roy J, Burke MD. Synthesis of most polyene natural product motifs using just 12 building blocks and one coupling reaction. Nat Chem. 2014 Jun;6(6):484-91. doi: 10.1038/nchem.1947. PMID 24848233
- [Background] Yang YL, Xiang ZJ, Yang JH, Wang WJ, Xu ZC, Xiang RL. Adverse Effects Associated With Currently Commonly Used Antifungal Agents: A Network Meta-Analysis and Systematic Review. Front Pharmacol. 2021 Oct 29;12:697330. doi: 10.3389/fphar.2021.697330. eCollection 2021. PMID 34776941
- [Background] Yoshida M, Tamura K, Masaoka T, Nakajo E. A real-world prospective observational study on the efficacy and safety of liposomal amphotericin B in 426 patients with persistent neutropenia and fever. J Infect Chemother. 2021 Feb;27(2):277-283. doi: 10.1016/j.jiac.2020.10.005. Epub 2020 Oct 24. PMID 33109439
- [Background] Zarakas MA, Desai JV, Chamilos G, Lionakis MS. Fungal Infections with Ibrutinib and Other Small-Molecule Kinase Inhibitors. Curr Fungal Infect Rep. 2019 Sep;13(3):86-98. doi: 10.1007/s12281-019-00343-9. Epub 2019 Jul 5. PMID 31555394
- [Background] Zhang Y, Holland E, Dinh A, Au D, Sun L. Bombesin-drug conjugates in targeted therapy for small cell lung cancer. Am J Cancer Res. 2022 Mar 15;12(3):927-937. eCollection 2022. PMID 35411251